CLINICAL TRIAL: NCT02354261
Title: Phase IIb Open-label Trial of SUBA™-Itraconazole in Subjects With Basal Cell Carcinoma Nevus Syndrome (BCCNS)
Brief Title: Open-label Trial of SUBA™-Itraconazole (SUBA-Cap) in Subjects With Basal Cell Carcinoma Nevus Syndrome (BCCNS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HedgePath Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP2001; SCORING (Other: HedgePath)
Record Dates: First submitted 2015-01-21; First posted 2015-02-03 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Basal Cell Carcinoma in Basal Cell Nevus Syndrome
Keywords: Basal Cell Carcinoma Nevus Syndrome; BCCNS; BCC; itraconazole; basal cell carcinoma; locally advanced basal cell carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SUBA-Itraconazole (Experimental): Subjects will receive an oral dose of 300 mg SUBA-itraconazole daily.
  Interventions: Drug: SUBA-Itraconazole

INTERVENTIONS:
Drug: SUBA-Itraconazole — Subjects will receive an oral dose of 300 mg SUBA-Itraconazole daily.
  Other Names: SUBA-Cap

SUMMARY:
The study will assess the safety and efficacy of SUBA-Cap in subjects with Basal Cell Carcinoma Nevus Syndrome.

DETAILED DESCRIPTION:
Single arm, phase IIb, multi-center, open-label study evaluating the use of oral SUBA-Cap in subjects with Basal Cell Carcinoma Nevus Syndrome and non-metastatic Basal Cell Carcinoma.

Following informed consent, subjects will undergo a skin biopsy for Gli1 analysis and an assessment of extent of disease using both tumor measurements (using modified Response Evaluation Criteria in Solid Tumors criteria) and color photographs of the skin.

Subjects will receive daily oral SUBA-Cap, at a starting dose of 150 mg twice daily (BID). Reassessments of disease will be conducted at weeks 4, 8, 16, and then every 8 weeks thereafter. Subjects with evidence of response (partial or complete) will be re-evaluated at least 4 weeks later for confirmation. Subjects may continue to receive SUBA-Cap until disease progression (defined as the appearance of one or more new lesions or ulceration of a target lesion) that requires a change in therapy (surgical intervention or use of other systemic therapy) or the appearance of unacceptable side effects. Pharmacokinetic assessments (serial trough levels) will be performed at defined intervals and, when possible, prior to and following any dose adjustment. Skin biopsies will be taken for Gli1 expression at defined intervals.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0 or 1
* Diagnosis of Basal Cell Carcinoma Nevus Syndrome (BCCNS)
* Histologic confirmation of BCC from at least one lesion
* History of surgical removal of at least ten (10) prior BCCs
* Measurable disease as defined, namely at least ten (10) measurable lesions such that the sum of the longest diameters of the measurable lesions is at least 40 mm.
* Has failed, refused, or is not eligible for standard of care therapy for BCC
* Willingness to abstain from the use of non-study treatments for BCC, including but not limited to topical medications, PDT, and/or irradiation therapy.
* At least four weeks from prior major surgery
* Women who are pre-menopausal or not surgically sterile must be willing to use an acceptable contraceptive method for the duration of the study and for 30 days following the last dose of study drug
* Sexually active men must be willing to use an acceptable contraceptive method for the duration of time on study and for 30 days following the last dose of study drug
* Clinical laboratory values within the following ranges:

  1. Negative serum pregnancy test
  2. Adequate hematologic function (ANC ≥1.5 x 10^9/L; platelet count ≥75x10^9/L; hemoglobin ≥9g/dL (in the absence of red blood cell transfusions in the prior 14 days)
  3. Prothrombin time (PT-INR) or activated partial thromboplastin time (APTT) <1.5 times the upper limit of normal range, unless currently receiving anticoagulants
  4. Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥60 mL/min
  5. Total bilirubin ≤ 1.5x the upper limit of normal unless considered due to Gilbert syndrome in which case, ≤ 3x the upper limit of normal
  6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels ≤ the upper limit of normal
* Willingness to undergo biopsies (BCC lesions and normal skin)
* Willingness to provide prior and study-related BCC biopsies for central review
* Willingness to participate in collection of pharmacokinetic samples
* Willingness to not donate blood, semen, or eggs for the duration of the study and for 3 months following discontinuation of SUBA-Cap
* Willingness to delay removal of otherwise surgically eligible BCC's

Exclusion Criteria:

* Presence of metastatic BCC
* Subjects who would be disserved significantly by a delay in conventional therapy, such as surgical intervention of their BCC
* Prior use of a hedgehog inhibitor (e.g., sonidegib, vismodegib) or Itraconazole within the past 6 months
* History of progressive disease on a hedgehog inhibitor (e.g., sonidegib, vismodegib) or other Hh pathway inhibitors for the treatment of BCC
* Pregnant and/or nursing women
* Use of any medications metabolized by the cytochrome P450 3A4 isoenzyme system (CYP3A4) known to lead to potentially serious and/or life threatening adverse events when used in conjunction with itraconazole
* Any illness that is likely to reduce absorption of oral medications
* Corrected QT (Fridericia) interval of >450 msec for females and >430 msec for males
* Use of any medications known to result in a prolongation of the QT interval
* History of congestive heart failure or other cardiac abnormality that would contraindicate the use of itraconazole
* Any condition or situation which in the Investigator's opinion may put the subject at significant risk, could confound the study results, or could interfere significantly with the subject's participation in the study
* Any indication of compromised liver function that would otherwise contraindicate use of itraconazole
* Any concurrent malignancy, except for squamous cell carcinoma of the skin and cervical carcinoma in situ, that is likely to require treatment within the next two years or would interfere with study requirements
* Psychiatric illness and/or social situations (e.g., excessive alcohol use or use of illicit drugs) that would interfere with study compliance
* Known HIV infection, active hepatitis B or active hepatitis C infection (testing not required unless indicated by history)
* Known allergy to itraconazole or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Response rate of BCC lesions | Up to 26 weeks

SECONDARY OUTCOMES:
Safety and tolerance; measured by number of subjects with adverse events | Participants will be followed for the duration of study participation, an expected average of 26 weeks
Number of new BCCs eligible for surgical resection | Up to 26 weeks
Duration of response in those subjects that have responded | Up to 26 weeks
Time to next therapy (systemic therapy or surgical intervention) | Up to 26 weeks
Change in the number of jaw cysts | Up to 26 weeks
Changes in the number of palmar/plantar pits | Up to 26 weeks
Gli1 expression in normal skin | Up to 26 weeks
Levels of itraconazole and hydroxy-itraconazole in the skin | Up to 26 weeks
Levels of itraconazole and hydroxy-itraconazole in the blood | For Cycle 1 and Cycle 2, Up to week 8

CONTACTS AND LOCATIONS:
Overall Officials: James Solomon, MD, PhD, Principal Investigator — Ameriderm Clinical Research
Locations (5):
- United States (5):
  - Dermatology Specialists, Inc, Oceanside, California
  - Ameriderm Research, Ormond Beach, Florida
  - Grekin Skin Institute, Warren, Michigan
  - Stony Brook University, East Setauket, New York
  - Penn State Hershey Medical Center, Hershey, Pennsylvania